CLINICAL TRIAL: NCT07346547
Title: Registry of Daprodustat in Chronic Kidney Disease (CKD) Anemia for Understanding Real-World Evidence (REDCURE)
Brief Title: REDCURE Registry for Chronic Kidney Disease (CKD) Anemia
Acronym: REDCURE
Status: Not yet recruiting | Type: Observational
Sponsor: Nabiqasim Industries (Pvt) Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NQ/DP/JES/Reg-006
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: CKD Anemia
Keywords: Daprodustat; oral HIF PHI; CKD anemia
MeSH Terms: interventions — GSK1278863

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Daprodustat arm for CKD anemia patients: Daprodustat arm for CKD anemia patients
  Interventions: Drug: Daprodustat

INTERVENTIONS:
Drug: Daprodustat — Hypoxia Inducible Factor (HIF) Prolyl Hydroxylase Inhibitor (PHI) drug

SUMMARY:
A local registry on CKD-associated anemia aims to provide real-world insights into disease burden, treatment patterns, and outcomes at the national level. It helps capture variations in anemia severity with CKD stages, therapeutic practices and their response. It also supports evidence-based decision-making, identifies gaps in care, and informs locally relevant guidelines and policy planning to improve patient outcomes with oral novel therapy i.e. daprodustat

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years 2. Diagnosed CKD-associated anemia Chronic Kidney Disease (CKD) diagnosed as per KDIGO criteria, including: CKD stages G3-G5 (based on eGFR)

  * Patients on hemodialysis (HD) or peritoneal dialysis (PD)
  * Post-kidney transplant patients with CKD 3. Receiving or initiating Daprodustat therapy (new start or switch therapy) 4. CKD stages 3-5, dialysis patients (HD/PD), or post-transplant with CKD anemia 5. Able and willing to provide informed consent

Exclusion Criteria

1. Acute Kidney Injury (AKI) without underlying chronicity
2. Hematologic disorders not related to CKD (e.g hemolytic anemia, aplastic anemia)
3. Refusal or inability to provide consent
4. Current enrollment in an interventional trial that restricts real-world data collection
5. Life expectancy < 3 months, where follow-up is not feasible
6. Known contraindications to Daprodustat as per local prescribing information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Chronic Kidney Disease (CKD) anemia requiring anemia treatment
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Serum hemoglobin levels | 3 months
  Hemoglobin response to therapy

SECONDARY OUTCOMES:
Frequency of MACE ( Major Adverse Cardiovascular Events) | 3 months
  MACE events:
  * Unstable angina requiring hospitalization
  * Non-fatal MI
  * Non-fatal stroke
  * Cardiovascular death
    * Other adverse events
    * Hospitalization episodes
      . Mortality
    * Optional patient-reported outcomes (fatigue, functional status)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0158765
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31582227/
- See also: Related Info — https://journals.plos.org/plosone/article?id=10.1371/journal.pone.0084943
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30352554/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25102850/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40937334/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30360959/